CLINICAL TRIAL: NCT04390126
Title: COVID-19 Related Lockdown Effects On Chronic Diseases
Acronym: CLEO-CD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BOULIN AOIc 2020
Record Dates: First submitted 2020-05-14; First posted 2020-05-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Chronic Coronary Syndrome; Heart Failure; AMD and Macular Edema; Chronic Respiratory Failure; Hemophilia; Malignant Hemopathy; Multiple Sclerosis; Horton's Disease
MeSH Terms: conditions — Heart Failure; Macular Edema; Hemophilia A; Multiple Sclerosis; Giant Cell Arteritis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Register of haematological malignancies
  Interventions: Other: life questionnaires; Other: questionnaire
- Idiopathic Pulmonary Fibrosis and PAH Cohort
  Interventions: Other: life questionnaires; Other: questionnaire
- Giant Cell Arteritis Cohort
  Interventions: Other: life questionnaires; Other: questionnaire
- AMD and Macular Edema Cohort
  Interventions: Other: life questionnaires; Other: questionnaire
- Multiple Sclerosis Cohort
  Interventions: Other: life questionnaires; Other: questionnaire
- Myocardial Infarction Observatory RICO
  Interventions: Other: life questionnaires; Other: questionnaire
- Heart Failure Cohort
  Interventions: Other: life questionnaires; Other: questionnaire
- Hemophilia Cohort
  Interventions: Other: life questionnaires; Other: questionnaire

INTERVENTIONS:
Other: life questionnaires — Telephone survey during the confinement period (common questionnaire and a questionnaire specific to the patient's pathology)
Other: questionnaire — 1-year telephone diary to identify complications resulting in hospitalization related to the patient's chronic disease

SUMMARY:
The containment associated with the VIDOC-19 pandemic creates an unprecedented societal situation of physical and social isolation. Our hypothesis is that in patients with chronic diseases, confinement leads to changes in health behaviours, adherence to pharmacological treatment, lifestyle rules and increased psychosocial stress with an increased risk of deterioration in their health status in the short, medium and long term.

Some messages about the additional risk/danger associated with taking certain drugs in the event of COVID disease have been widely disseminated in the media since March 17, 2020, the date on which containment began in France. This is the case, for example, for corticosteroids, non-steroidal anti-inflammatory drugs but also for converting enzyme inhibitors (ACE inhibitors) and angiotensin II receptor antagonists (ARBs2). These four major classes of drugs are widely prescribed in patients with chronic diseases, diseases specifically selected in our study (corticosteroids: haematological malignancies, multiple sclerosis, Horton's disease; ACE inhibitors/ARAs2: heart failure, chronic coronary artery disease). Aspirin used at low doses as an anti-platelet agent in coronary patients as a secondary prophylaxis after a myocardial infarction can be stopped by some patients who consider aspirin to be a non-steroidal anti-inflammatory drug. Discontinuation of this antiplatelet agent, which must be taken for life after an infarction, exposes the patient to a major risk of a new cardiovascular event.

The current difficulty of access to care due to travel restrictions (a theoretical limit in the context of French confinement but a priori very real), the impossibility of consulting overloaded doctors, or the cancellation of medical appointments, medical and surgical procedures due to the reorganization of our hospital and private health system to better manage COVID-19 patients also increases the risk of worsening the health status of chronic patients who by definition require regular medical monitoring.

Eight Burgundian cohorts of patients with chronic diseases (chronic coronary artery disease, heart failure, multiple sclerosis, Horton's disease, AMD, haemopathic malignancy, chronic respiratory failure (idiopathic fibrosis, PAH) haemophilia cohort) will study the health impact of the containment related to the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* patients with one of the following chronic diseases: chronic coronary syndrome, heart failure, multiple sclerosis, Horton's disease, AMD, malignant haemopathy, chronic respiratory failure (idiopathic fibrosis, PAH, haemophilia) and already registered in one of the 8 Burgundian registries/cohorts.

Exclusion Criteria:

* deceased patient, patient cannot be reached after >3 telephone calls, patient or caregiver does not speak French to carry out telephone interviews

Min Age: 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients from existing registries or cohorts
Sampling Method: Non-Probability Sample
Enrollment: 1343 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
% adherence to each pharmacological class | during the period from 20 April 2020 to 7 May 2020
  increase in dose, decrease in dose, discontinuation or no change for each drug class)
number of occurrence of medical events at 1 year | throughout the study for 12 months
  (mortality, hospitalizations and relevant criteria for each pathology all related to the chronic disease)

SECONDARY OUTCOMES:
Expressed in %: Non-pharmacological treatment/lifestyle: | during the period from 20 April 2020 to 7 May 2020
  Smoking/Smoking/sweetening, Alcohol consumption/recovery, Decreased physical activity, Weight change
Expressed in %: Difficulties accessing care: medical appointments, prescriptions, medication | during the period from 20 April 2020 to 7 May 2020
Measurement of psychological distress: Kessler's specific questionnaire (score between 0 and 24) | during the period from 20 April 2020 to 7 May 2020

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Boulin M, Cransac-Miet A, Maynadie M, Volot F, Creuzot-Garcher C, Eicher JC, Chague F, Ksiazek E, Beltramo G, Bonniaud P, Moreau T, Bonnotte B, Sales-Wuillemin E, Soudry-Faure A, Zeller M, Cottin Y. COVID-19 Lockdown in Patients with Chronic Diseases: A Cross-Sectional Study. Int J Environ Res Public Health. 2022 Mar 26;19(7):3957. doi: 10.3390/ijerph19073957. PMID 35409640
- [Derived] Volot F, Soudry-Faure A, Callegarin A, Ksiazek E, Delienne S, Cottin Y, Maynadie M, Boulin M. Impact of first COVID-19 lockdown on paediatric and adult haemophilia patients treated in a French Haemophilia Comprehensive Care Centre. Haemophilia. 2022 May;28(3):462-471. doi: 10.1111/hae.14526. Epub 2022 Mar 3. PMID 35238436